CLINICAL TRIAL: NCT00941512
Title: Investigation to Correlate High Resolution Digital Images of the Uterine Cervix With Histopathology
Brief Title: High Resolution Digital Imaging of the Uterine Cervix
Status: Completed | Type: Observational
Sponsor: STI-Medical Systems (Industry)
Collaborators: Instituto National de Edfermedades Neoplasicas (Unknown); Eisenhower Army Medical Center (U.S. Federal Agency)
Responsible Party: Jody Oyama, STI Medical Systems
Other Study IDs: 2005-1
Record Dates: First submitted 2009-07-15; First posted 2009-07-17 (Estimated); Last update posted 2009-07-17 (Estimated); Status verified 2009-07

CONDITIONS: Colposcopy
Keywords: Colposcopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Uterine Cervix tissue
Oversight: Data Monitoring Committee: No

SUMMARY:
This study was designed to gather digital pictures of the cervix and correlate it to its histopathology, and then use those relationships to teach a computer how to objectively find cervical dysplasia and cancer.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Negative pregnancy test
* 18 years and older
* Presence of a cervix

Exclusion Criteria:

* Pregnant
* Absence of a cervix
* Less than 18 years old
* Male

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women identified with an abnormal Pap smear
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2005-04; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daron G Ferris, Principal Investigator — Augusta University